CLINICAL TRIAL: NCT00385710
Title: Randomized Placebo-controlled Trial of Valproic Acid in Patients With Progressive Supranuclear Palsy
Brief Title: Trial of Valproic Acid in Patients With Progressive Supranuclear Palsy (Depakine)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/10-H
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2011-05

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive supranuclear palsy (PSP)
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- valproic acid (Experimental): Depakine
  Interventions: Drug: valproic acid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: valproic acid — Depakine
  Arms: valproic acid
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Progressive Supranuclear Palsy (PSP) is a relentlessly progressive neurodegenerative disorder, clinically characterized by parkinsonism with prominent axial involvement and postural instability, bulbar symptoms, supranuclear ophthalmoplegia, and executive dysfunction. Abnormal neuronal and glial tau aggregations affecting the basal ganglia and selective brainstem structures result in dysfunction of the five frontosubcortical circuits and brainstem functions. There is no effective treatment for PSP. One of the key feature in the aggregation of tau is its phosphorylation by kinases such as glycogen synthase kinase 3b (GSK3b). Recent reports have shown that valproic acid was able to inhibit the activity of GSK3b and could exert a neuroprotective effect through this inhibition. The investigators thus decided to conduct this controlled study to assess the putative neuroprotective effects in patients with PSP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with possible or probable PSP
* from 45 to 75 year of age

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
PSPRS score (specific score for PSP) | This score will be measured every three months during the two-year follow up of the study

SECONDARY OUTCOMES:
Neuropsychological evaluation | inclusion, one year and two years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Derkinderen, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - Service de Neurologie A, Hôpital Gabriel Montpied-BP, Clermont-Ferrand
  - Service de Neurologie et Pathologie du mouvement Hôpital Roger Salingro, CHRU de Lille, Lille
  - Service de Neurologie, CHU Nantes, Nantes
  - Service de Neurologie, CHU Poitiers, Poitiers